CLINICAL TRIAL: NCT02519361
Title: The Involvement of the Translation Initiation Factors eIF4E and eIF4G in Resolution of Inflammation in the Elderly Population
Brief Title: Involvement of the Translation Initiation Factors in Resolution of Inflammation in the Elderly Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0148-15-MMC
Record Dates: First submitted 2015-08-02; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Infection in the Elderly
Keywords: elderly; immune response; acute infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aging cause specific changes in the immune system. Processes like "immunoessence" and "inflammaging" offend the functioning of the immune cells and expose the elderly patient to infections that can lead to morbidity and death.

Protein translation regulation offers a strategic advantage to the immune cells, because it enables rapid activation or termination of synthesis of specific proteins, required for inflammation or its resolution. Translation initiation depends on recruitment of eukaryotic initiation factor "eIF4F" complex.

The aim of the current study is to investigate the involvement of the translation initiation factors (eIF4E and eIF4G) in the process of recovery from acute infection in elderly patient admitted to the internal department with an acute infection.

DETAILED DESCRIPTION:
1. Blood samples of elderly patients diagnosed with acute infection (fever and leukocytosis) will be collected twice - at admittance to Meir hospital and after recovery (24-48 hours without fever and leukocytosis). evidence of infection (chest x ray, urine and blood samples) will be collected. participants will be divided to two age groups: 65-80 yrs and very old patient >85 yrs, and will be compared to younger patients aged 50-65.
2. Peripheral blood samples will be separated to subpopulations of lymphocytes, monocytes and polymorphonuclears, and protein will be extracted.
3. protein lysates will be separated by SDS-PAGE electrophoresis and immunoblotted for phosphorylated and total eIF4E and eIF4G; their regulators: Mnk 1/2, 4EBP1, mTOR and targets: cyclin D1, c-Myc, survivin, BCL2, VEGFA, etc.
4. Paired samples (within each age group) will be analyzed and correlated with clinical response of the patients. The source of the infection will also be considered.
5. Comparison between age groups at admittance and upon recovery will be made (Unpaired).

ELIGIBILITY:
Inclusion Criteria:

* patient aged 50 y and more with:
* fever >38c that started in the 48 hours prior to admission
* leukocytosis >10.0 K/microLiter
* suspected source of infection by symptoms, lab results or imaging
* treatment with antibiotics started in the last 24 hours or is about to be started

Exclusion Criteria:

* patients who cannot sign the informed concent ( dementia)
* patients with active malignancy
* patients who are under chemotherapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to internal department due to acute infection
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Translation initiation factors expression by immunoblotting, in leukocytes sub population | 1 week
  Assessment of eIF4E and eIF4G expression by immunoblotting, in leukocytes sub populations under inflamed conditions and upon resolution of acute inflammation, in three groups of age

SECONDARY OUTCOMES:
Translation initiation factors regulators expression by immunoblotting in leukocytes sub population | 1 week
  Assessment of eIF4E and eIF4G regulators expression by immunoblotting, in leukocytes sub populations under inflamed conditions and upon resolution of acute inflammation in three age groups
Translation initiation factors targets expression by immunoblotting in leukocytes sub population | 1 week
  Assessment of eIF4E and eIF4G targets expression by immunoblotting in leukocytes sub populations under inflamed conditions and upon resolution of acute inflammation, in three age groups

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Heffez Ayzenfeld, MD, Principal Investigator — r.h.ayzenfeld